CLINICAL TRIAL: NCT07133958
Title: A Bidirectional Observational Clinical Study of Tumor Regression Patterns in Patients With Locally Advanced Oral and Oropharyngeal Squamous Cell Carcinoma Treated With Neoadjuvant Immunochemotherapy
Brief Title: A Bidirectional Observational Clinical Study of NAIC in the Treatment of Tumor Regression Patterns in LA-OSCC and LA-OPSCC
Status: Recruiting | Type: Observational
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-KY-195
Record Dates: First submitted 2025-08-14; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Oral Squamous Cell Carcinoma (OSCC); Oropharyngeal Squamous Cell Carcinoma (SCC)
Keywords: Oral squamous cell carcinoma; Oropharyngeal squamous cell carcinoma; neoadjuvant immunochemotherapy
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A prospective collection of 35 cases was conducted at Zhujiang Hospital of Southern Medical University. Patients diagnosed with locally advanced oral squamous cell carcinoma (LA-OSCC) or locally advanced oropharyngeal squamous cell carcinoma (LA-OPSCC) from April 2023 onward, who received two cycles of neoadjuvant immunochemotherapy (tislelizumab + paclitaxel + cisplatin/carboplatin) at our institution, were included. The study analyzed treatment safety, efficacy, tumor regression patterns, 2-year progression-free survival (PFS), and 5-year overall survival (OS) rates.

DETAILED DESCRIPTION:
This study retrospectively collected data from patients in 2023 and prospectively collected data from patients undergoing treatment at the same time. In terms of time type, it is a bidirectional study. Meanwhile, these studies are a single-arm, single-center study and belong to a case series study.

ELIGIBILITY:
Inclusion Criteria:

1. Oral squamous cell carcinoma or oropharyngeal squamous cell carcinoma diagnosed as locally advanced (T3-4) according to the AJCC criteria
2. Their age ranged from 18 to 80 years
3. There was no history of other malignant tumors or treatment
4. Adequate blood function: white blood cell count (WBC) ≥3.5×10^9/L, platelet count (PLT) ≥75×10^9/L; Hemoglobin concentration (HGB) ≥90g/L
5. Adequate liver function: total bilirubin (TBIL) ≤ the upper limit of normal, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 times the upper limit of normal
6. "Adequate renal function: urinary white blood cells < 10, red blood cells < 10, cast count < 5 per high-power field, and creatinine (CRE) ≤ the upper limit of normal.
7. The heart, brain, lung and other vital organs function and general condition can tolerate NACI and surgical treatment
8. PS score ≤2

Exclusion Criteria:

1. Presence of distant metastasis
2. Women who are pregnant or lactating
3. Patients who are unable to cooperate with regular follow-up due to psychological, social, family and geographical reasons
4. Receiving investigational treatment in addition to other clinical studies (in the treatment phase of a clinical study)
5. Accompanied by severe uncontrolled infection or medical illness
6. Major organ dysfunction, such as decompensated heart, lung, kidney, and liver failure, cannot tolerate NACI or surgical treatment
7. There are factors affecting surgery or anesthesia, such as severe organ dysfunction
8. Long-term use of immunosuppressive agents after organ transplantation
9. Patients with a history of other malignant tumors before enrollment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants were planned to receive 2 cycles of intravenous neoadjuvant Tislelizumab (200 mg) every 3 weeks,and Paclitaxel 135-175mg/m2, Cisplatin 80-120mg/m2 or Carboplatin 0.3-0.4g/m2 through intravenous infusion each 3-week cycle for 2cycles.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2023-07-11 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
0bjective Response Rate | 8 weeks
  According to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. it isdefined as the proportion of patients who achieved Complete Response (CR) or Partial Response(PR).Complete Response (CR) was defined as disappearance of all target lesions. PartialResponse (PR) was defined as >=30% decrease in the sum of the longest diameter of targetlesions.

SECONDARY OUTCOMES:
Tumor regression pattern | 8 weeks
  ①Concentric Shrinkage Mode (CS): Refers to a unified inward contraction of tumor cells toward the lesion center as a cohesive unit, without residual scattered tumor foci at the periphery.
  ②Non-Concentric Shrinkage Mode (NCS): Also termed "Dendritic Shrinkage" or "Nest-like/Marginal Shrinkage", characterized by: Heterogeneous regression of the tumor mass, manifesting as: a) Fragmentation of the primary lesion into discontinuous satellite nodules, OR b) Preservation of the original tumor dimensions with heterogeneously reduced density.
two-year progression-free survival rate | 2 years
  The proportion of patients who remain alive and progression-free for 2 years aftertreatment

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Stomatology, Zhujiang Hospital, Southern Medical University,Guangzhou, Guangdong, Guangzhou, Guangdong, China